CLINICAL TRIAL: NCT02452931
Title: An Open-label, Single Arm, Multicenter Study on the Efficacy, Safety, and Pharmacokinetics of Leuprolide Acetate 45 mg for Injectable Suspension Controlled Release in Subjects With Central (Gonadotropin-Dependent) Precocious Puberty
Brief Title: Study of Leuprolide Acetate Injectable Suspension in the Treatment of Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tolmar Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOL2581A; NCT02811471 (obsolete NCT alias)
Record Dates: First submitted 2015-05-05; First posted 2015-05-25 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Precocious Puberty, Central
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Assigned Intervention (Experimental): Leuprolide acetate 45 mg will be administered as a subcutaneous injection at 6-month intervals for the 12 month study period.
  Interventions: Drug: Leuprolide Acetate 45 mg

INTERVENTIONS:
Drug: Leuprolide Acetate 45 mg — Subcutaneous injection

SUMMARY:
This study determines the effectiveness of leuprolide acetate 45 mg for injectable suspension for treatment of children with Central Precocious Puberty.

DETAILED DESCRIPTION:
Leuprolide acetate is a GnRH agonist that inhibits pituitary gonadotropin secretion by binding to the GnRH receptors and blocking downstream hormone synthesis. The steady decrease in hormone synthesis (LH and FSH) leads to a suppression of testicular and ovarian steroidogenesis. In children with CPP, this steady decrease in hormone synthesis disrupts the progression of puberty.

ELIGIBILITY:
Inclusion Criteria:

* Females age 2 to 8 years (inclusive) or males age 2 to 9 years (inclusive)
* Confirmed diagnosis of CPP within 12 months of Baseline Visit (Day 0) but have not received prior GnRH agonist treatment for CPP
* Pubertal-type LH response following an abbreviated GnRHa stimulation test before treatment initiation
* Clinical evidence of puberty, defined as Tanner stage ≥ 2 for breast development in females or testicular volume ≥ 4 mL in males
* Difference between bone age (Greulich and Pyle method) and chronological age ≥ 1 year

Exclusion Criteria:

* Gonadotropin-independent (peripheral) precocious puberty
* Prior or current GnRH treatment for CPP
* Prior or current therapy with medroxyprogesterone acetate, growth hormone or insulin-like growth factor-1 (IGF-1)
* Diagnosis of short stature (ie, 2.25 standard deviations (SD) below the mean height for age)
* Known history of seizures, epilepsy, and/or central nervous system disorders that may be associated with seizures or convulsions
* Any other medical condition or serious intercurrent illness that, in the opinion of the Investigator, may make it undesirable for the subject to participate in the study

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Schorr, Study Director — orphan reach USA, LLC
Locations (20):
- United States (10):
  - University of California, San Diego, San Diego, California
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Endocrine, Cincinnati, Ohio
  - University of Oklahoma College of Medicine, Tulsa, Oklahoma
  - Seattle Children's, Seattle, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
- Hospital de Ninos, Buenos Aires, Argentina
- Canada (3):
  - University of Calgary, Alberta Children's Hospital, Calgary, Alberta
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec
- Chile (3):
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Instituto de Investigaciones Materno Infantil (IDIMI), Santiago, Santiago Metropolitan
  - Hospital Regional de Antofagasta Leonardo Guzman, Antofagasta, Second Region
- Mexico (2):
  - Hospital Unversitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Instituto de Investigaciones Aplicadas a la Neurociencia, A.C., Durango
- The Liggins Institute, University of Auckland, Auckland, New Zealand

REFERENCES:
- [Derived] Klein KO, Freire A, Gryngarten MG, Kletter GB, Benson M, Miller BS, Dajani TS, Eugster EA, Mauras N. Phase 3 Trial of a Small-volume Subcutaneous 6-Month Duration Leuprolide Acetate Treatment for Central Precocious Puberty. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3660-71. doi: 10.1210/clinem/dgaa479. PMID 32738042

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Assigned Intervention
Started | 64
Completed | 60
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (0.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 3
  Black or African American | 15
  Native Hawaiian or Other Pacific Islander | 1
  White | 34
  Unwilling to Provide | 1
  Other | 5
  Hispanic or Latino | 36
  Not hispanic or Latino | 28
Region of Enrollment [Number; unit: participants]
  New Zealand | 2
  Canada | 2
  Argentina | 13
  United States | 31
  Mexico | 7
  Chile | 9
Luteinizing Hormone [Mean (Standard Deviation); unit: IU/L] — Pubertal-type LH response following an abbreviated GnRHa stimulation test before treatment initiation > 5 IU/L Population: The Overall number of participants represents the Safety population. The Study analysis used the Intent-to-Treat (ITT) population: Subjects providing consent/assent who received at least one dose of the study drug, fulfilled the protocol eligibility criteria, and provided at least one PD laboratory assessment post dosing.
  IU/L
    number analyzed (Participants) | 62
    (all) | 23.46 (24.282)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of Peak-Stimulated Luteinizing Hormone at 6 Months.
Description: Luteinizing Hormone (LH) suppression is defined as peak-stimulated LH <4 IU/L. Peak stimulated LH refers to the maximum LH concentration measured 30 minutes after a gonadotropin-releasing hormone agonst (GnRHa) stimulation test.
Time Frame: 6 months
Population: Intent-to-Treat (ITT) population: Subjects providing consent/assent who received at least one dose of the study drug, fulfilled the protocol eligibility criteria, and provided at least one PD laboratory assessment post dosing.
Measure: Count of Participants; unit: Participants
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Participants | 54

2. Secondary Outcome: Percentage of Subjects With Suppression of Luteinizing Hormone Measured by Blood Levels.
Description: Percentage of subjects with suppressed serum LH concentrations(<4 IU/L) 30 minutes post GnRHa stimulation test at all assessed timepoints.
Time Frame: Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Participants
  Visit 3, Week 12: number analyzed (Participants) | 60
  Visit 3, Week 12 | 51
  Visit 5, Week 24 | 54
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 50
  End of Treatment, Week 48: number analyzed (Participants) | 58
  End of Treatment, Week 48 | 50

3. Secondary Outcome: Changes in Height Velocity (Growth Rate)
Description: Changes in height velocity (growth rate) at all study timepoints after Screening to end of study. Growth velocity is defined for each visit as change from baseline / [(number of weeks since baseline)/52]. Week 48: Change from Week 24 growth velocity is defined as change from week 24 to week 48 / [(number of weeks since week 24)/52].
Time Frame: Week 4, Week 12, Week 20, Week 24, Week 36, Week 44, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
cm/year
  Visit 2, Week 4 | 8.89 (13.128)
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12 | 8.30 (4.782)
  Visit 4, Week 20: number analyzed (Participants) | 60
  Visit 4, Week 20 | 6.66 (3.155)
  Visit 5, Week 24: number analyzed (Participants) | 61
  Visit 5, Week 24 | 6.90 (3.074)
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 6.48 (2.272)
  Visit 7, Week 44: number analyzed (Participants) | 59
  Visit 7, Week 44 | 6.23 (1.953)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 6.37 (1.893)
  End of Treatment, Week 48: Change from Week 24: number analyzed (Participants) | 59
  End of Treatment, Week 48: Change from Week 24 | 5.79 (2.213)

4. Secondary Outcome: Bone Age Ratio to Chronological Age at Time of Measurement
Description: Bone Age Ratio to Chronological Age at Time of Measurement is bone age/age at bone age assessment.
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Ratio
  Baseline | 1.39 (0.160)
  Visit 5, Week 24 | 1.34 (0.138)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 1.32 (0.143)
  Minimum Post-baseline Value | 1.30 (0.138)
  Maximum Post-baseline Value | 1.36 (0.138)

5. Secondary Outcome: Percent Change From Baseline in Height
Description: The percent change from baseline in height at each available post-baseline measurement. Percent change is defined as (((change from Baseline)/(Baseline)) x 100).
Time Frame: Week 4, Week 12, Week 20, Week 24, Week 36, Week 44, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Percent change
  Visit 2, Week 4 | 0.5 (0.78)
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12 | 1.4 (0.82)
  Visit 4, Week 20: number analyzed (Participants) | 60
  Visit 4, Week 20 | 1.9 (0.89)
  Visit 5, Week 24: number analyzed (Participants) | 61
  Visit 5, Week 24 | 2.3 (1.06)
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 3.3 (1.17)
  Visit 7, Week 44: number analyzed (Participants) | 59
  Visit 7, Week 44 | 3.9 (1.26)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 4.3 (1.34)

6. Secondary Outcome: Tanner Scores: Boys - Development of External Genitalia
Description: Sexual development (physical signs) in puberty were assessed by Tanner staging, a system developed by Marshall and Tanner to categorize pubertal maturation. Tanner stages are commonly used to categorize pubertal maturation in terms of sequence, timing and tempo. Tanner Stages: the minimum is Stage 1 = pre-pubertal physical characteristics and the maximum is Stage 5 = fully matured (adult) physical characteristics.
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 2
Score on a scale
  Baseline | 3.0 (0.00)
  Visit 3, Week 12 | 2.5 (0.71)
  Visit 5, Week 24 | 2.5 (0.71)
  Visit 6, Week 36 | 2.5 (0.71)
  End of Treatment, Week 48 | 2.0 (0.00)

7. Secondary Outcome: Tanner Scores: Boys - Development of External Genitalia (Change From Baseline)
Description: as for outcome 6
Time Frame: Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 2
Score on a scale
  Visit 3, Week 12 | -0.5 (0.71)
  Visit 5, Week 24 | -0.5 (0.71)
  Visit 6, Week 36 | -0.5 (0.71)
  End of Treatment, Week 48 | -1.0 (0.00)

8. Secondary Outcome: Tanner Scores: Boys and Girls - Pubic Hair
Description: as for outcome 6
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Score on a scale
  Baseline | 2.3 (0.81)
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12 | 2.4 (0.89)
  Visit 5, Week 24 | 2.5 (0.92)
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 2.3 (0.94)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 2.4 (0.95)

9. Secondary Outcome: Tanner Scores: Boys and Girls - Pubic Hair (Change From Baseline)
Description: as for outcome 6
Time Frame: Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Score on a scale
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12 | 0.1 (0.56)
  Visit 5, Week 24 | 0.1 (0.59)
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 0.1 (0.60)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 0.1 (0.58)

10. Secondary Outcome: Tanner Scores: Girls - Breast Development
Description: as for outcome 6
Time Frame: Baseline, Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 60
Score on a scale
  Baseline | 3.2 (0.61)
  Visit 3, Week 12: number analyzed (Participants) | 59
  Visit 3, Week 12 | 2.7 (0.90)
  Visit 5, Week 24 | 2.6 (1.0)
  Visit 6, Week 36: number analyzed (Participants) | 57
  Visit 6, Week 36 | 2.5 (0.89)
  End of Treatment, Week 48: number analyzed (Participants) | 57
  End of Treatment, Week 48 | 2.4 (0.93)

11. Secondary Outcome: Tanner Scores: Girls - Breast Development (Change From Baseline)
Description: as for outcome 6
Time Frame: Week 12, Week 24, Week 36, and Week 48
Population: Intent-to-Treat (ITT) population: Subjects providing consent/assent who received at least one dose of the study drug, fulfilled the protocol eligibility criteria, and provided at least one PD laboratory assessment post dosing. Tanner Stages: I (<10yrs), II (10-11yrs), III (11-13yrs), IV (13-14yrs), V (>14yrs).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 60
Score on a scale
  Visit 3, Week 12: number analyzed (Participants) | 59
  Visit 3, Week 12 | -0.5 (0.90)
  Visit 5, Week 24 | -0.6 (0.87)
  Visit 6, Week 36: number analyzed (Participants) | 57
  Visit 6, Week 36 | -0.6 (0.86)
  End of Treatment, Week 48: number analyzed (Participants) | 57
  End of Treatment, Week 48 | -0.7 (0.89)

12. Other Pre Specified Outcome: Height
Description: Height at each available measurement point. Baseline is defined as the last non-missing height measurement collected prior to or on the date of first injection.
Time Frame: Screening, Baseline, Week 4, Week 12, Week 20, Week 24, Week 36, Week 44, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
cm
  Screening | 136.17 (8.292)
  Baseline | 136.61 (8.071)
  Visit 2, Week 4 | 137.32 (8.201)
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12 | 138.52 (8.284)
  Visit 4, Week 20: number analyzed (Participants) | 60
  Visit 4, Week 20 | 138.87 (8.070)
  Visit 5, Week 24: number analyzed (Participants) | 61
  Visit 5, Week 24 | 139.78 (8.206)
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36 | 140.99 (8.374)
  Visit 7, Week 44: number analyzed (Participants) | 59
  Visit 7, Week 44 | 141.81 (8.268)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 142.37 (8.207)

13. Other Pre Specified Outcome: Bone Age
Description: Bone Age at each available measurement point.
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
years
  Baseline | 11.01 (1.307)
  Visit 5, Week 24 | 11.30 (1.238)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 11.65 (1.124)

14. Other Pre Specified Outcome: Bone Age Progression
Description: Bone age progression at each available post-baseline measurement point. Bone age progression is defined as (((change from baseline)/(baseline)) x 100), which is percent change from baseline.
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
percent change
  Visit 5, Week 24 | 2.91 (4.607)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 6.81 (5.741)
  Minimum Post-Baseline Value | 2.91 (4.607)
  Maximum Post-Baseline Value | 6.63 (5.736)

15. Other Pre Specified Outcome: Bone Age Ratio to Chronological Age at Time of Measurement (Percent Change From Baseline)
Description: Bone Age Ratio to Chronological Age at Time of Measurement is bone age/age at bone age assessment.
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
percent change
  Visit 5, Week 24 | -3.25 (4.382)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | -4.90 (4.689)
  Minimum Post-baseline Value | -6.15 (3.934)
  Maximum Post-baseline Value | -1.89 (4.155)

16. Other Pre Specified Outcome: Bone Age Ratio to Chronological Age at Start of Study (Percent Change From Baseline)
Description: Bone age advancement was evaluated relative to chronological age at each given measurement point. Percent change from baseline is: 100 x (the change from baseline value at the post-baseline visit / baseline value).
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
percent change
  Visit 5, Week 24 | 2.91 (4.607)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 6.81 (5.741)
  Minimum Post-baseline Value | 2.91 (4.607)
  Maximum Post-baseline Value | 6.63 (5.736)

17. Other Pre Specified Outcome: Bone Age Ratio to Chronological Age at Start of Study
Description: Bone age advancement was evaluated relative to chronological age at each given measurement point. Bone Age Ratio to Chronological Age at Start of Study is bone age/age at first injection.
Time Frame: Baseline, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Ratio
  Baseline | 1.38 (0.158)
  Visit 5, Week 24 | 1.42 (0.153)
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48 | 1.47 (0.178)
  Minimum Post-baseline Value | 1.42 (0.153)
  Maximum Post-baseline Value | 1.47 (0.176)

18. Other Pre Specified Outcome: GnRH Antagonist Evaluation
Description: GnRH Antagonist Evaluation occurred for the two week period following each treatment and at each visit to assess flare symptoms. The percent of subjects who affirm (or whose parent/guardian affirms) each symptom domain in the global interview.
Time Frame: Week 2, Week 4, Week 12, Week 20, Week 24, Week 26, Week 36, Week 44, and Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Participants
  Telephone Contact #1, Week 2: number analyzed (Participants) | 59
  Telephone Contact #1, Week 2: Any GnRH Antagonist Conditions Reported? | 15
  Telephone Contact #1, Week 2: Flare or hot flashes | 4
  Telephone Contact #1, Week 2: Injection site reactions | 11
  Telephone Contact #1, Week 2: Burning/Stinging | 0
  Telephone Contact #1, Week 2: Pain | 9
  Telephone Contact #1, Week 2: Bruising | 3
  Telephone Contact #1, Week 2: Redness | 0
  Telephone Contact #1, Week 2: Difficulty in urination | 1
  Telephone Contact #1, Week 2: Bone Pain | 1
  Telephone Contact #1, Week 2: Aggravation of weakness or other muscle symptoms | 0
  Telephone Contact #1, Week 2: Onset of Allergic reactions | 0
  Telephone Contact #1, Week 2: No GnRH Antagonist conditions reported? | 15
  Visit 2, Week 4: Any GnRH Antagonist Conditions Reported? | 4
  Visit 2, Week 4: Flare or hot flashes | 2
  Visit 2, Week 4: Injection site reactions | 1
  Visit 2, Week 4: Burning/Stinging | 0
  Visit 2, Week 4: Pain | 1
  Visit 2, Week 4: Bruising | 0
  Visit 2, Week 4: Redness | 0
  Visit 2, Week 4: Difficulty in urination | 0
  Visit 2, Week 4: Bone Pain | 1
  Visit 2, Week 4: Aggravation of weakness or other muscle symptoms | 0
  Visit 2, Week 4: Onset of Allergic reactions | 0
  Visit 2, Week 4: No GnRH Antagonist conditions reported? | 53
  Visit 3, Week 12: number analyzed (Participants) | 61
  Visit 3, Week 12: Any GnRH Antagonist Conditions Reported? | 5
  Visit 3, Week 12: Flare or hot flashes | 1
  Visit 3, Week 12: Injection site reactions | 3
  Visit 3, Week 12: Burning/Stinging | 0
  Visit 3, Week 12: Pain | 2
  Visit 3, Week 12: Bruising | 0
  Visit 3, Week 12: Redness | 1
  Visit 3, Week 12: Difficulty in urination | 0
  Visit 3, Week 12: Bone Pain | 1
  Visit 3, Week 12: Aggravation of weakness or other muscle symptoms | 0
  Visit 3, Week 12: Onset of Allergic reactions | 0
  Visit 3, Week 12: No GnRH Antagonist conditions reported? | 48
  Visit 4, Week 20: number analyzed (Participants) | 60
  Visit 4, Week 20: Any GnRH Antagonist Conditions Reported? | 3
  Visit 4, Week 20: Flare or hot flashes | 1
  Visit 4, Week 20: Injection site reactions | 1
  Visit 4, Week 20: Burning/Stinging | 0
  Visit 4, Week 20: Pain | 1
  Visit 4, Week 20: Bruising | 0
  Visit 4, Week 20: Redness | 0
  Visit 4, Week 20: Difficulty in urination | 0
  Visit 4, Week 20: Bone Pain | 1
  Visit 4, Week 20: Aggravation of weakness or other muscle symptoms | 0
  Visit 4, Week 20: Onset of Allergic reactions | 0
  Visit 4, Week 20: No GnRH Antagonist conditions reported? | 53
  Visit 5, Week 24: number analyzed (Participants) | 61
  Visit 5, Week 24: Any GnRH Antagonist Conditions Reported? | 3
  Visit 5, Week 24: Flare or hot flashes | 1
  Visit 5, Week 24: Injection site reactions | 1
  Visit 5, Week 24: Burning/Stinging | 0
  Visit 5, Week 24: Pain | 0
  Visit 5, Week 24: Bruising | 0
  Visit 5, Week 24: Redness | 0
  Visit 5, Week 24: Difficulty in urination | 0
  Visit 5, Week 24: Bone Pain | 1
  Visit 5, Week 24: Aggravation of weakness or other muscle symptoms | 0
  Visit 5, Week 24: Onset of Allergic reactions | 0
  Visit 5, Week 24: No GnRH Antagonist conditions reported? | 55
  Telephone Contact #2, Week 26: number analyzed (Participants) | 57
  Telephone Contact #2, Week 26: Any GnRH Antagonist Conditions Reported? | 16
  Telephone Contact #2, Week 26: Flare or hot flashes | 2
  Telephone Contact #2, Week 26: Injection site reactions | 15
  Telephone Contact #2, Week 26: Burning/Stinging | 0
  Telephone Contact #2, Week 26: Pain | 15
  Telephone Contact #2, Week 26: Bruising | 0
  Telephone Contact #2, Week 26: Redness | 3
  Telephone Contact #2, Week 26: Difficulty in urination | 0
  Telephone Contact #2, Week 26: Bone Pain | 0
  Telephone Contact #2, Week 26: Aggravation of weakness or other muscle symptoms | 0
  Telephone Contact #2, Week 26: Onset of Allergic reactions | 0
  Telephone Contact #2, Week 26: No GnRH Antagonist conditions reported? | 6
  Visit 6, Week 36: number analyzed (Participants) | 59
  Visit 6, Week 36: Any GnRH Antagonist Conditions Reported? | 3
  Visit 6, Week 36: Flare or hot flashes | 1
  Visit 6, Week 36: Injection site reactions | 1
  Visit 6, Week 36: Burning/Stinging | 0
  Visit 6, Week 36: Pain | 1
  Visit 6, Week 36: Bruising | 0
  Visit 6, Week 36: Redness | 1
  Visit 6, Week 36: Difficulty in urination | 1
  Visit 6, Week 36: Bone Pain | 0
  Visit 6, Week 36: Aggravation of weakness or other muscle symptoms | 0
  Visit 6, Week 36: Onset of Allergic reactions | 0
  Visit 6, Week 36: No GnRH Antagonist conditions reported? | 51
  Visit 7, Week 44: number analyzed (Participants) | 59
  Visit 7, Week 44: Any GnRH Antagonist Conditions Reported? | 3
  Visit 7, Week 44: Flare or hot flashes | 2
  Visit 7, Week 44: Injection site reactions | 0
  Visit 7, Week 44: Burning/Stinging | 0
  Visit 7, Week 44: Pain | 0
  Visit 7, Week 44: Bruising | 0
  Visit 7, Week 44: Redness | 0
  Visit 7, Week 44: Difficulty in urination | 0
  Visit 7, Week 44: Bone Pain | 0
  Visit 7, Week 44: Aggravation of weakness or other muscle symptoms | 0
  Visit 7, Week 44: Onset of Allergic reactions | 1
  Visit 7, Week 44: No GnRH Antagonist conditions reported? | 53
  End of Treatment, Week 48: number analyzed (Participants) | 59
  End of Treatment, Week 48: Any GnRH Antagonist Conditions Reported? | 1
  End of Treatment, Week 48: Flare or hot flashes | 1
  End of Treatment, Week 48: Injection site reactions | 0
  End of Treatment, Week 48: Burning/Stinging | 0
  End of Treatment, Week 48: Pain | 0
  End of Treatment, Week 48: Bruising | 0
  End of Treatment, Week 48: Redness | 0
  End of Treatment, Week 48: Difficulty in urination | 0
  End of Treatment, Week 48: Bone Pain | 0
  End of Treatment, Week 48: Aggravation of weakness or other muscle symptoms | 0
  End of Treatment, Week 48: Onset of Allergic reactions | 0
  End of Treatment, Week 48: No GnRH Antagonist conditions reported? | 57

19. Other Pre Specified Outcome: Percentage of Subjects With Suppression of FSH, Estradiol, Oestradiol (HS), and Testosterone Measured by Blood Levels.
Description: The percentage of subjects with FSH, estradiol and testosterone suppression to prepubertal levels (FSH < 2.5 mIU/mL, estradiol < 20 pg/mL and testosterone < 28.4 ng/dL) at each available time point.
Time Frame: Week 12, Week 24, Week 36, and Week 48
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Participants
  Visit 3, Week 12 : FSH: number analyzed (Participants) | 60
  Visit 3, Week 12 : FSH | 37
  Visit 3, Week 12 : Estradiol: number analyzed (Participants) | 58
  Visit 3, Week 12 : Estradiol | 58
  Visit 3, Week 12 : Oestradiol (HS): number analyzed (Participants) | 57
  Visit 3, Week 12 : Oestradiol (HS) | 56
  Visit 3, Week 12 : Testosterone: number analyzed (Participants) | 2
  Visit 3, Week 12 : Testosterone | 2
  Visit 5, Week 24 : FSH | 41
  Visit 5, Week 24 : Estradiol: number analyzed (Participants) | 60
  Visit 5, Week 24 : Estradiol | 59
  Visit 5, Week 24 : Oestradiol (HS): number analyzed (Participants) | 60
  Visit 5, Week 24 : Oestradiol (HS) | 58
  Visit 5, Week 24 : Testosterone: number analyzed (Participants) | 2
  Visit 5, Week 24 : Testosterone | 2
  Visit 6, Week 36 : FSH: number analyzed (Participants) | 59
  Visit 6, Week 36 : FSH | 26
  Visit 6, Week 36 : Estradiol: number analyzed (Participants) | 57
  Visit 6, Week 36 : Estradiol | 57
  Visit 6, Week 36 : Oestradiol (HS): number analyzed (Participants) | 57
  Visit 6, Week 36 : Oestradiol (HS) | 56
  Visit 6, Week 36 : Testosterone: number analyzed (Participants) | 2
  Visit 6, Week 36 : Testosterone | 2
  End of Treatment, Week 48 : FSH: number analyzed (Participants) | 58
  End of Treatment, Week 48 : FSH | 32
  End of Treatment, Week 48 : Estradiol: number analyzed (Participants) | 56
  End of Treatment, Week 48 : Estradiol | 56
  End of Treatment, Week 48 : Oestradiol (HS): number analyzed (Participants) | 56
  End of Treatment, Week 48 : Oestradiol (HS) | 55
  End of Treatment, Week 48 : Testosterone: number analyzed (Participants) | 2
  End of Treatment, Week 48 : Testosterone | 1

20. Other Pre Specified Outcome: Changes in the Ratio of LH/FSH
Description: Changes in ratio of LH/FSH at each time point from Screening to End of Study
Time Frame: Screening (Pre&Post GnRHa Stim Test), Baseline (0,1,4,6 hours Post-Injection), Week 4, Week 12 (Pre&Post GnRHa Stim Test), Week 20, Week 24 (Pre&Post GnRHa Stim Test), Week 36 (Pre&Post GnRHa Stim Test), Week 44, and Week 48 (Pre&Post GnRHa Stim Test)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Assigned Intervention
Number analyzed (Participants) | 62
Ratio
  Screening: Pre GnRHa Stimulation Test | 0.387 (0.4675)
  Screening: Post GnRHa Stimulation Test: number analyzed (Participants) | 61
  Screening: Post GnRHa Stimulation Test | 2.187 (1.6713)
  Baseline | 0.604 (0.9851)
  Baseline: 1 hr Post Inj: number analyzed (Participants) | 60
  Baseline: 1 hr Post Inj | 2.424 (2.1534)
  Baseline: 1 hr Post Inj: Change from Baseline: number analyzed (Participants) | 60
  Baseline: 1 hr Post Inj: Change from Baseline | 1.856 (1.7277)
  Baseline: 4 hr Post Inj: number analyzed (Participants) | 60
  Baseline: 4 hr Post Inj | 2.110 (2.3939)
  Baseline: 4 hr Post Inj: Change from Baseline: number analyzed (Participants) | 60
  Baseline: 4 hr Post Inj: Change from Baseline | 1.542 (2.0932)
  Baseline: 6 hr Post Inj: number analyzed (Participants) | 60
  Baseline: 6 hr Post Inj | 1.691 (1.7330)
  Baseline: 6 hr Post Inj: Change from Baseline: number analyzed (Participants) | 60
  Baseline: 6 hr Post Inj: Change from Baseline | 1.123 (1.4378)
  Week 4: number analyzed (Participants) | 60
  Week 4 | 0.843 (1.0004)
  Week 4: Change from Baseline: number analyzed (Participants) | 60
  Week 4: Change from Baseline | 0.233 (1.1425)
  Week 12: Pre GnRHa Stim Test: number analyzed (Participants) | 60
  Week 12: Pre GnRHa Stim Test | 0.565 (0.9100)
  Week 12: Pre GnRHa Stim Test: Change from Baseline: number analyzed (Participants) | 60
  Week 12: Pre GnRHa Stim Test: Change from Baseline | -0.050 (1.0423)
  Week 12: Post GnRHa Stim Test: number analyzed (Participants) | 60
  Week 12: Post GnRHa Stim Test | 1.342 (1.7934)
  Week12: Post GnRHa Stim Test: Change from Baseline: number analyzed (Participants) | 60
  Week12: Post GnRHa Stim Test: Change from Baseline | 0.721 (1.7237)
  Week 20: number analyzed (Participants) | 59
  Week 20 | 0.654 (0.9806)
  Week 20: Change from Baseline: number analyzed (Participants) | 59
  Week 20: Change from Baseline | 0.068 (1.1859)
  Week 24: Pre GnRHa Stim Test | 0.611 (0.9571)
  Week 24: Pre GnRHa Stim Test: Change from Baseline | 0.007 (1.1818)
  Week 24: Post GnRHa Stim Test | 1.320 (1.2843)
  Week24: Post GnRHa Stim Test: Change from Baseline | 0.716 (1.4450)
  Week 36: Pre GnRHa Stim Test: number analyzed (Participants) | 58
  Week 36: Pre GnRHa Stim Test | 0.474 (0.5249)
  Week 36: Pre GnRHa Stim Test: Change from Baseline: number analyzed (Participants) | 58
  Week 36: Pre GnRHa Stim Test: Change from Baseline | -0.125 (1.0038)
  Week 36: Post GnRHa Stim Test: number analyzed (Participants) | 59
  Week 36: Post GnRHa Stim Test | 1.051 (1.4130)
  Week36: Post GnRHa Stim Test: Change from Baseline: number analyzed (Participants) | 59
  Week36: Post GnRHa Stim Test: Change from Baseline | 0.461 (15374)
  Week 44: number analyzed (Participants) | 59
  Week 44 | 0.517 (0.7846)
  Week 44: Change from Baseline: number analyzed (Participants) | 59
  Week 44: Change from Baseline | -0.073 (1.0575)
  Week 48: Pre GnRHa Stim Test: number analyzed (Participants) | 59
  Week 48: Pre GnRHa Stim Test | 0.557 (1.0957)
  Week 48: Pre GnRHa Stim Test: Change from Baseline: number analyzed (Participants) | 59
  Week 48: Pre GnRHa Stim Test: Change from Baseline | -0.033 (1.2191)
  Week 48: Post GnRHa Stim Test: number analyzed (Participants) | 58
  Week 48: Post GnRHa Stim Test | 1.092 (1.5655)
  Week48: Post GnRHa Stim Test: Change from Baselin: number analyzed (Participants) | 58
  Week48: Post GnRHa Stim Test: Change from Baselin | 0.509 (1.5780)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time ICF was signed until End of Treatment (48 weeks). Any AEs related to study drug were followed for 28 days or through resolution, stabilization, until deemed clinically insignificant, or until the subject is lost to follow-up.
Description: Definition of Suspected Adverse Reaction is any AE for which there is reasonable possibility that the drug caused the AE. Definition of Unexpected Adverse Event is an AE or suspected adverse reaction considered unexpected if it is not listed in the ELIGARD® Package Insert, or is not listed in the Investigator Brochure.
Arm/Group | Assigned Intervention
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 1/64
Other Adverse Events (participants affected / at risk) | 55/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assigned Intervention (N=64)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Assigned Intervention (N=64)
Abdominal pain (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Pyrexia (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 14
Upper respiratory tract infection (Infections and infestations) | 4
Headache (Nervous system disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protocol Section 11.3 Publication, the Investigator shall not make any publication related to this study without the express written permission of the Sponsor. The Investigator agrees to provide abstract, manuscript, and/or documentation for Sponsor review 90 days prior to submission for publication/presentation. The Sponsor retains the right to delete from the manuscript confidential information and to object to suggested publication and/or its timing (at the Sponsor's sole discretion).

DOCUMENTS (2):
  • Study Protocol (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT02452931/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02452931/SAP_001.pdf